CLINICAL TRIAL: NCT06647888
Title: A Multi-Center, Observational Study to Evaluate the Efficacy and Safety of Enavogliflozin in Patients With Type II Diabetes Mellitus Accompanied by Hypertension or Dyslipidemia
Brief Title: Evaluation of Enavogliflozin's Efficacy and Safety in Type II Diabetes With Hypertension or Dyslipidemia
Status: Recruiting | Type: Observational
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Other Study IDs: DWENV_DB_02
Record Dates: First submitted 2024-10-16; First posted 2024-10-18 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Enavogliflozin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Envlo Tablet — Envlo Tab. 0.3mg
  Other Names: Enavogliflozin 0.3mg
Drug: Envlomet SR Tablet — Envlomet SR Tablet 0.3/ Metformin1,000mg
  Other Names: Enavogliflozin 0.3mg/ Metformin1,000mg

SUMMARY:
This observational study is a non-interventional, multi-center, prospective observational study aimed at tracking the efficacy and safety of Envlo or Envlomet SR tablets for 24 weeks in patients with type 2 diabetes and hypertension or dyslipidemia who are currently taking or are scheduled to take Envlo or Envlomet SR tablets in an actual clinical setting.

DETAILED DESCRIPTION:
This observational study planned recruit population of type 2 diabetes patients who are scheduled to administer Envlo tablet or Envlomet SR Tablet according to the medical judgment of the researcher (doctor in charge) based on permission (efficacy & effect, usage & dose, usage precautions, etc.) in the actual treatment environment.

This observational study will be conducted in an actual treatment environment regardless of whether Envlo tablet or Envlomet SR Tablet was administered or not.

Information such as demographic information, body measurement, and vital signs performed will be collected up to 24 weeks after Envlo tablet or Envlomet SR Tablet administration.

Data will be collected based on medical records recorded in the actual treatment environment, and there is no mandatory visit, examination, or treatment in this observation study.

ELIGIBILITY:
Inclusion Criteria:

1. An adult male and female over 19 years of age
2. A patient diagnosed with type 2 diabetes who have hypertension or dyslipidemia and are currently receiving Envlo Tab/ Envlomet SR Tab or are scheduled to receive Envlo Tab/ Envlomet SR Tab
3. A person who voluntarily participates in the observational study and agrees in writing to comply with the subject's precautions during the study period after hearing and understanding the detailed explanation of the characteristics of the observational study and the drug to be studied 4 ) A person who understands the content of this observational study, are cooperative with the research process, and are considered capable of participating until the study's completion

Exclusion Criteria:

1. Among patients who begin treatment with Envlo Tab/ Envlomet Tab at the time of registration, those with an estimated glomerular filtration rate (eGFR) of less than 60 ml/min/1.73m²
2. A patient with diabetes other than type 2 diabetes (type 1 diabetes, diabetic ketoacidosis, gestational diabetes, etc.)
3. A person who is prohibited from administering in accordance with the permission of Envlo Tab's

   * Patients who overreact to Envlo Tab or Envlomet Tab components and have a history of it
   * Patients with an estimated glomerular filtration rate (eGFR) of less than 60 ml/min/1.73m², end-stage renal disease, or on dialysis
   * Patients with moderate and severe liver failure (AST or ALT > 3x normal upper limit, Total Bilirubin > 2x normal upper limit, hepatitis or liver failure)
   * Class III or IV by classification of the New York Heart Association (NYHA)
4. Patients with unstable weight due to treatment or other treatments (surgery, diet, etc.) with obesity or weight loss medication within 3 months of Enrollment
5. Pregnant women and lactating women
6. A person who participates in another clinical trial and is administering (applying) clinical trial drugs or clinical trial medical devices
7. A person who is considered inappropriate to participate in this observational study based on the judgment of investigators

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The proportion of study participants reaching the target blood glucose levels of HbA1c < 7.0% or FPG < 126 mg/dL at the 24-week mark compared to baseline was estimated using PASS 14. The minimum number of participants required to generate a two-sided 95% confidence interval is calculated to be 9,604. Considering an approximate dropout rate of 25%, we plan to recruit a total of 12,000 study participants.
Sampling Method: Non-Probability Sample
Enrollment: 12000 (Estimated)
Dates: Start 2024-12-03 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Target achievement rates for blood glucose | at 24 weeks
  Target achievement rates for blood glucose at 24 weeks
Target achievement rates for LDL-C treatment goals | at 24 weeks
  Target achievement rates for LDL-C treatment goals at 24 weeks
Target control rates for blood pressure | at 24 weeks
  Target control rates for blood pressure at 24 weeks

SECONDARY OUTCOMES:
change in HbA1c | 12 week
  change in HbA1c at 12 week compared to baseline
change in HbA1c | 24 week
  change in HbA1c at 24 week compared to baseline
change in FPG | 12 week
  change in FPG at 12 week compared to baseline
change in FPG | 24 week
  change in FPG at 24 week compared to baseline
percentage of subjects achieved HbA1c < 7 % | 12 week
  percentage of subjects achieved HbA1c < 7 % at 12 week compared to baseline
percentage of subjects achieved HbA1c < 7 % | 24 week
  percentage of subjects achieved HbA1c < 7 % at 24 week compared to baseline
percentage of subjects achieved HbA1c < 6.5 % | 12 week
  percentage of subjects achieved HbA1c < 6.5 % at 12 week compared to baseline
percentage of subjects achieved HbA1c < 6.5 % | 24 week
  percentage of subjects achieved HbA1c < 6.5 % at 24 week compared to baseline
therapeutic response(change in HbA1c > 0.5 % OR HbA1c < 7 %) | 12 week
  therapeutic response(change in HbA1c > 0.5 % OR HbA1c < 7 %) at 12 week compared to baseline
therapeutic response(change in HbA1c > 0.5 % OR HbA1c < 7 %) | at 24 week
  therapeutic response(change in HbA1c > 0.5 % OR HbA1c < 7 %) at 24 week compared to baseline
change in blood pressure (systolic blood pressure, diastolic blood pressure) | at 12 week
  change in blood pressure (systolic blood pressure, diastolic blood pressure) at 12 week compared to baseline
change in blood pressure (systolic blood pressure, diastolic blood pressure) | at 24 week
  change in blood pressure (systolic blood pressure, diastolic blood pressure) at 24 week compared to baseline
change in lipid profiles (Total Cholesterol, LDL-C, HDL-C, Triglyceride) | at 12 week
  change in lipid profiles (Total Cholesterol, LDL-C, HDL-C, Triglyceride) at 12 week compared to baseline
change in lipid profiles (Total Cholesterol, LDL-C, HDL-C, Triglyceride) | at 24 week
  change in lipid profiles (Total Cholesterol, LDL-C, HDL-C, Triglyceride) at 24 week compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Sang Hoon Moon, Principal Investigator — Happy Yonsei Family Medicine Clinic
Locations (1):
- Happy Yonsei Family Medicine Clinic, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided